CLINICAL TRIAL: NCT03068975
Title: A Double Blind, Randomized, Parallel Design Study to Evaluate the Effectiveness of Post-operative Dose of Alvimopan(Entereg) in Preventing Post-operative Ileus in Poly-traumatized Patients
Brief Title: Alvimopan Use in Polytraumatized Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated due to failure to enroll, a low volume of patients met criteria.
Sponsor: University of Puerto Rico (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pablo Rodriguez Ortiz, MD, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 55238
Record Dates: First submitted 2017-02-17; First posted 2017-03-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Post Operative Ileus
MeSH Terms: interventions — alvimopan

STUDY DESIGN:
Intervention Model Description: Will create a double blind, randomized, parallel design study to evaluate the effectiveness of Alvimopan(post operative dose) in preventing post-operative ileus in poly-traumatized patients
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alvimopan (Experimental): Patients in the study group will be administered a post operative dose of Alvimopan
  Interventions: Drug: Alvimopan
- Placebo (Placebo Comparator): Patients in the Placebo group will receive a placebo pill and will be compared with the study group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — Patients who sustained abdominal trauma with resection of bowel and anastomosis will receive Alvimopan ( post operative dose only) and will monitor for post operative ileus.
  Other Names: Entereg
  Arms: Alvimopan
Drug: Placebo — Patients who sustained abdominal trauma with resection of bowel and anastomosis will receive the Placebo Pill (post operative dose only) and will monitor for post operative ileus.
  Other Names: placebo pill
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of Alvimopan(12 mg) in recovery of bowel function in an emergency trauma setting without the pre-operative dosage in patients that will receive abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 80
* Poly-traumatized patients
* Extubated patients after abdominal exploration
* Underwent Abdominal exploration, had colon resection with primary anastomosis with closure of abdomen

Exclusion Criteria:

* Mechanically ventilated patients
* Patient not expected to survive Glasgow Coma Scale = 3
* Pregnant patients
* Apache score > 40 (observed mortality 100%) Saas Ahmed Naved et al 2011
* Vasopressor therapy
* Septic patients
* Thoracotomy
* Bogota bag
* Intravenous Drug Abuser (IVDA) as evidenced by urine toxicology upon admission to the Trauma Unit
* Patients with prior history of gastric surgery and/or colonic surgery
* Medical History: of severe cardiovascular disease, Renal diseases, Hepatitis C or Hepatic failure, Autoimmune disease, Crohn and Ulcerative Colitis (In view of the inflammation in the intestinal mucosal which may decrease optimal absorption of the medication) and or bowel obstruction
* Prior pancreatic anastomosis or gastric anastomosis; ostomy formation
* Chronic use of nonsteroidal anti-inflammatory drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Recovery of bowel function in trauma patients who received post operative dose of Alvimopan compared to placebo. | 2 years
  Since Entereg is a peripherally opioid receptor antagonist it will bind to those receptors and will avoid the post operative ileus hence the bowel recovery will be faster. By physical examination (passage of flatus, bowel movements upon auscultation) will be used to assess recovery of bowel function

SECONDARY OUTCOMES:
Length of stay in patients of the same population who receive a placebo. | 5 years
  Since Entereg is a peripherally opioid receptor antagonist it will bind to those receptors and will avoid the post operative ileus and all the associated complications that prolonged the length of stay of the patients, hence it will reduce the hospital days of the individual

CONTACTS AND LOCATIONS:
Locations (1):
- Puerto Rico Trauma Hospital, San Juan, US, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bragg D, El-Sharkawy AM, Psaltis E, Maxwell-Armstrong CA, Lobo DN. Postoperative ileus: Recent developments in pathophysiology and management. Clin Nutr. 2015 Jun;34(3):367-76. doi: 10.1016/j.clnu.2015.01.016. Epub 2015 Jan 31. PMID 25819420
- [Background] Delaney CP, Weese JL, Hyman NH, Bauer J, Techner L, Gabriel K, Du W, Schmidt WK, Wallin BA; Alvimopan Postoperative Ileus Study Group. Phase III trial of alvimopan, a novel, peripherally acting, mu opioid antagonist, for postoperative ileus after major abdominal surgery. Dis Colon Rectum. 2005 Jun;48(6):1114-25; discussion 1125-6; author reply 1127-9. doi: 10.1007/s10350-005-0035-7. PMID 15906123
- [Background] Delaney CP, Senagore AJ, Viscusi ER, Wolff BG, Fort J, Du W, Techner L, Wallin B. Postoperative upper and lower gastrointestinal recovery and gastrointestinal morbidity in patients undergoing bowel resection: pooled analysis of placebo data from 3 randomized controlled trials. Am J Surg. 2006 Mar;191(3):315-9. doi: 10.1016/j.amjsurg.2005.10.026. PMID 16490538
- [Background] Earnshaw SR, Kauf TL, McDade C, Potashman MH, Pauyo C, Reese ES, Senagore A. Economic Impact of Alvimopan Considering Varying Definitions of Postoperative Ileus. J Am Coll Surg. 2015 Nov;221(5):941-50. doi: 10.1016/j.jamcollsurg.2015.08.004. Epub 2015 Aug 15. PMID 26353904
- [Background] Hilton WM, Lotan Y, Parekh DJ, Basler JW, Svatek RS. Alvimopan for prevention of postoperative paralytic ileus in radical cystectomy patients: a cost-effectiveness analysis. BJU Int. 2013 Jun;111(7):1054-60. doi: 10.1111/j.1464-410X.2012.11499.x. Epub 2012 Nov 21. PMID 23171223
- [Background] Herzog TJ, Coleman RL, Guerrieri JP Jr, Gabriel K, Du W, Techner L, Fort JG, Wallin B. A double-blind, randomized, placebo-controlled phase III study of the safety of alvimopan in patients who undergo simple total abdominal hysterectomy. Am J Obstet Gynecol. 2006 Aug;195(2):445-53. doi: 10.1016/j.ajog.2006.01.039. Epub 2006 Apr 19. PMID 16626607
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Kalff JC, Schraut WH, Simmons RL, Bauer AJ. Surgical manipulation of the gut elicits an intestinal muscularis inflammatory response resulting in postsurgical ileus. Ann Surg. 1998 Nov;228(5):652-63. doi: 10.1097/00000658-199811000-00004. PMID 9833803
- [Background] Ludwig K, Viscusi ER, Wolff BG, Delaney CP, Senagore A, Techner L. Alvimopan for the management of postoperative ileus after bowel resection: characterization of clinical benefit by pooled responder analysis. World J Surg. 2010 Sep;34(9):2185-90. doi: 10.1007/s00268-010-0635-9. PMID 20526599
- [Background] Ludwig K, Enker WE, Delaney CP, Wolff BG, Du W, Fort JG, Cherubini M, Cucinotta J, Techner L. Gastrointestinal tract recovery in patients undergoing bowel resection: results of a randomized trial of alvimopan and placebo with a standardized accelerated postoperative care pathway. Arch Surg. 2008 Nov;143(11):1098-105. doi: 10.1001/archsurg.143.11.1098. PMID 19015469
- [Background] Manger JP, Nelson M, Blanchard S, Helo S, Conaway M, Krupski TL. Alvimopan: A cost-effective tool to decrease cystectomy length of stay. Cent European J Urol. 2014;67(4):335-41. doi: 10.5173/ceju.2014.04.art4. Epub 2014 Dec 5. PMID 25667750
- [Background] Miedema BW, Johnson JO. Methods for decreasing postoperative gut dysmotility. Lancet Oncol. 2003 Jun;4(6):365-72. doi: 10.1016/s1470-2045(03)01118-5. PMID 12788410
- [Background] Naved SA, Siddiqui S, Khan FH. APACHE-II score correlation with mortality and length of stay in an intensive care unit. J Coll Physicians Surg Pak. 2011 Jan;21(1):4-8. PMID 21276376
- [Background] Simorov A, Thompson J, Oleynikov D. Alvimopan reduces length of stay and costs in patients undergoing segmental colonic resections: results from multicenter national administrative database. Am J Surg. 2014 Dec;208(6):919-25; discussion 925. doi: 10.1016/j.amjsurg.2014.08.011. Epub 2014 Sep 22. PMID 25440479
- [Background] Thompson M, Magnuson B. Management of postoperative ileus. Orthopedics. 2012 Mar;35(3):213-7. doi: 10.3928/01477447-20120222-08. PMID 22385598
- [Background] Vaughan-Shaw PG, Fecher IC, Harris S, Knight JS. A meta-analysis of the effectiveness of the opioid receptor antagonist alvimopan in reducing hospital length of stay and time to GI recovery in patients enrolled in a standardized accelerated recovery program after abdominal surgery. Dis Colon Rectum. 2012 May;55(5):611-20. doi: 10.1097/DCR.0b013e318249fc78. PMID 22513441
- [Background] Winegar B, Cox M, Truelove D, Brock G, Scherrer N, Pass LA. Efficacy of alvimopan following bowel resection: a comparison of two dosing strategies. Ann Pharmacother. 2013 Nov;47(11):1406-13. doi: 10.1177/1060028013504289. PMID 24285757
- [Background] Wolff BG, Michelassi F, Gerkin TM, Techner L, Gabriel K, Du W, Wallin BA; Alvimopan Postoperative Ileus Study Group. Alvimopan, a novel, peripherally acting mu opioid antagonist: results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial of major abdominal surgery and postoperative ileus. Ann Surg. 2004 Oct;240(4):728-34; discussion 734-5. doi: 10.1097/01.sla.0000141158.27977.66. PMID 15383800